CLINICAL TRIAL: NCT01407900
Title: A Human Physiologic Study to Evaluate the Renal and Neurohumoral Effects of Dual NPR-A and NPR-B Activation With a Novel Chimeric Natriuretic Peptide (CD-NP)in Subjects With Stable Chronic Heart Failure and Moderate Renal Dysfunction
Brief Title: Effects of Chimeric Natriuretic Peptide Versus Placebo in Stable Heart Failure and Moderate Renal Dysfunction
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: New technique for administration of drug, this is the old technique of administration.
Sponsor: John A. Schirger (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, John A. Schirger, MD, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-008619
Record Dates: First submitted 2011-07-27; First posted 2011-08-02 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Heart Failure; Renal Insufficiency
Keywords: CD NP; dual receptor; NPR A; NPR B; Adult, aged over 45
MeSH Terms: conditions — Heart Failure; Renal Insufficiency | interventions — Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5% Dextrose in Water (Placebo Comparator): Infusion of D5W
  Interventions: Drug: 5% Dextrose in Water
- CD-NP (Active Comparator): CD-NP as a four hour infusion at 10 ng/kg/min IV
  Interventions: Drug: CD-NP

INTERVENTIONS:
Drug: CD-NP — CD-NP as a four hour infusion at 10 ng/kg/min IV
  Other Names: Chimeric natriuretic peptide
  Arms: CD-NP
Drug: 5% Dextrose in Water — four hour infusion IV
  Other Names: D5W
  Arms: 5% Dextrose in Water

SUMMARY:
The overall aim is to conduct a human physiologic study to assess the renal and neurohumoral effects of CD-NP vs placebo in older subjects with stable chronic systolic heart failure and moderate renal dysfunction.

DETAILED DESCRIPTION:
The investigators will evaluate the renal and neurohumoral effects of dual receptor (NPR-A and NPR-B) activation with CD-NP. This is a clinically relevant patient population who is at increased risk of developing diuretic resistance during the treatment of HF exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female with stable chronic HF of primary cardiac etiology, resting left ventricular ejection fraction (LVEF) ≤ 40 % documented within the last 2 years.
* Moderate renal dysfunction with creatinine clearance of 30-60 ml.min-1.1.73m-2, as calculated by Cockcroft-Gault formula24 and adjusted for body surface area within the past year or at screening, or requirement for dialysis.
* Be willing to provide informed consent.

Exclusion Criteria:

* Known allergy or other adverse reactions to exogenous natriuretic peptides (CD-NP or its components, nesiritide, other natriuretic peptides, or related compounds).
* Women who are pregnant, or breast-feeding, on hormonal contraceptives or hormone replacement therapy. (Women should be in the post-menopausal state, defined as the absence of menses for ≥ 1 year and serum follicle-stimulating hormone ≥ 20 IU/L; or should be previously sterilized defined as bilateral tubal occlusion for ≥ 6 months, bilateral oophorectomy, or complete hysterectomy)
* Having received nesiritide for within 7 days prior to prior to entry into the study.
* Having received any investigational drug or device within 30 days prior to entry into the study.
* Clinically unstable patients (e.g. systolic blood pressure < 90 mmHg, ongoing requirement for vasopressors or mechanical circulatory support, or mechanical ventilation).
* Recent hospitalization for decompensated HF or recent defibrillation for cardiac resuscitation within 30 days prior to randomization.
* Prior organ transplantation, being on a waiting list for organ transplantation, or ongoing requirement for long-term vasoactive support.
* Prior requirement for dialysis or ultrafiltration
* Active urinary tract infection
* Patients with guarded prognosis who are unlikely to derive meaningful benefit from CD-NP.
* Use of sulfonamides, non-steroidal anti-inflammatory drugs, probenecid, or other drugs that are known to alter renal function within one week of the first dose of CD-NP or placebo.
* Presence of cardiac lesions or comorbidities that may contraindicate the use of natriuretic peptides, such as clinically significant cardiac valvular stenosis, hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, or uncorrected congenital heart disease that contraindicates the use of vasodilators.
* History of blood pressure > 190/115 mmHg or unexplained syncope within the past 3 months.
* Symptomatic carotid artery disease, known critical carotid stenosis, or stroke within the past 3 months
* Clinically significant renal artery stenosis
* Baseline hemoglobin < 10.0 g/dl.
* Serum sodium < 130 mEq/L, potassium < 3.6 mEq/L, or magnesium < 1.7 mEq/L.
* Elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) at least 5 times the upper limit of normal or bilirubin at least 3 times the upper limit of normal
* History of alcohol abuse within the past 6 months.
* Consumption of a phosphodiesterase-5 inhibitor (sildenafil, vardenafil, or tadalafil) within 72 hours of receiving CD-NP or placebo.
* Inability to communicate effectively with study personnel.
* BMI >38

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in renal parameters | 1-hour period before drug or placebo infusion (baseline) and average of two 2-hour periods of drug or placebo infusion collected in a 5-hour period on the study day
  Renal parameters
  * Glomerular filtration rate, tubular function
  * Renal plasma flow
  * Urine output
  * Urinary sodium and potassium excretion
  * Urinary NGAL for early, acute alterations in renal function
  Change in value = [(Value during C2 + Value during C3)/2 ] - Value during C1
Change in hormonal parameters | 1-hour period before drug or placebo infusion (baseline) and average of two 2-hour periods of drug or placebo infusion collected in a 5-hour period on the study day
  Hormonal parameters
  * Plasma cyclic GMP, ANP, BNP, NT-proBNP, CNP, renin, angiotensin II, aldosterone, and norepinephrine
  * Urinary cyclic GMP, ANP, BNP, CNP
  * Plasma and urinary CD-NP
  Change in value = [(Value during C2 + Value during C3)/2 ] - Value during C1
Change in hemodynamic parameters | 1-hour period before drug or placebo infusion (baseline) and average of two 2-hour periods of drug or placebo infusion collected in a 5-hour period on the study day
  Hemodynamic parameters
  • Mean arterial pressure, heart rate
  Change in value = [(Value during C2 + Value during C3)/2 ] - Value during C1

CONTACTS AND LOCATIONS:
Overall Officials: John Schirger, MD, Principal Investigator — Mayo Clinic